CLINICAL TRIAL: NCT00669903
Title: A Phase IIa, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of Oral Multiple Ascending Doses of AZD0328 in Patients With Schizophrenia
Brief Title: Study to Asses Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of AZD0328 in Patients With Schizophrenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Since AZD0328 is unlikely to meet the current Target Product Profile, Astrazeneca decided to stop further development of AZD0328
Sponsor: AstraZeneca (Industry)
Responsible Party: Didier Meulien - Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D0190C00007
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Results first posted 2010-08-06 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — spiro(1-azabicyclo(2.2.2)octane-3,2'(3H)-furo(2,3-b)pyridine)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- 1 (Experimental): AZD0328 low dose
  Interventions: Drug: AZD0328
- 2 (Experimental): AZD0328 Optimal dose
  Interventions: Drug: AZD0328
- 3 (Experimental): AZD0328 High dose
  Interventions: Drug: AZD0328
- 4 (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD0328
  Arms: 1; 2; 3
Drug: Placebo
  Arms: 4

SUMMARY:
This study is to assess the pharmacodynamics, pharmacokinetics, safety and tolerability of multiple ascending doses of AZD0328 in patients with schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to the DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, 4th Edition)
* Low level of Extra-pyramidal symptoms
* No clinically significant findings on physical examination

Exclusion Criteria:

* Diagnosis of schizoaffective or schizophreniform disorders
* Any significant psychiatric or neurological disease other than schizophrenia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Center, Garden Grove, California
  - Research Center, Glendale, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of two US centers were inititated with first patient enrolled on 2 April 2008 and last patient completed on 4 November 2008. A total of 158 patients were enrolled with 100 patients allocated to randomized treatment.
Pre-assignment Details: Patients were to receive a stable dose of an antipsychotic for the 4 weeks prior to randomization, have stable psychotic symptoms without a hospitalization for the 8 weeks prior to randomization, and were to be smoking an average of >=10 cigarettes per day. Enrolled patients who no longer met entry criteria at randomization were not randomized.
Groups:
- AZD0328 Low Dose Group: AZD0328 Low dose group (0.00093 to 0.0028 mg oral solution)
- AZD0328 Optimal Dose Group: AZD0328 Optimal dose group (0.0048 to 0.0329 mg oral solution)
- AZD0328 High Dose Group: AZD0328 High dose group (0.075 to 0.675 mg oral solution)
- Placebo: Placebo
Period: Overall Study
Arm/Group | AZD0328 Low Dose Group | AZD0328 Optimal Dose Group | AZD0328 High Dose Group | Placebo
Started | 23 | 37 | 18 | 22
Completed Treatment Period | 23 | 33 | 13 | 19
Completed | 22 | 32 | 13 | 18
Not Completed | 1 | 5 | 5 | 4
Not completed — Adverse Event | 0 | 1 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD0328 Low Dose Group | AZD0328 Optimal Dose Group | AZD0328 High Dose Group | Placebo | Total
Number analyzed (Participants) | 23 | 37 | 18 | 22 | 100
Age Continuous [Mean (Standard Deviation); unit: Years] | 38.5 (11.2) | 41.7 (9.2) | 38.3 (9.8) | 40.0 (9.8) | 40.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 3 | 2 | 10
  Male | 22 | 33 | 15 | 20 | 90
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 4 | 3 | 1 | 2 | 10
  Black | 18 | 33 | 17 | 18 | 86
  Other | 1 | 1 | 0 | 2 | 4
Baseline Positive and Negative Syndrome Scale (PANSS) total score [Mean (Standard Deviation); unit: Points of PANSS score] — Baseline Positive and Negative Syndrome Scale (PANSS) total score. Best value for PANSS total score = 30 to worse value for PANSS total score = 210
  Points of PANSS score | 67.9 (10.3) | 71.8 (12.0) | 72.1 (12.2) | 69.5 (13.2) | 70.4 (11.9)

OUTCOME MEASURES:

1. Primary Outcome: CogState Groton Maze Learning Task (GMLT) and One Card Learning Task (OCLT) Standardized Composite Score at Day 14
Description: The GMLT and OCLT standardized change composite score will be calculated as the mean of the GMLT and OCLT standardized change from baseline scores. Least square means were derived using a mixed effects repeated measures model with protocol scheduled assessment day, treatment group, baseline score, and assessment day-by-treatment interaction as fixed factors, center as a random factor, and baseline score as a covariate. Scale range from negative infinity (worst value) to positive infinity (best value).
Time Frame: Baseline and Day 14
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZD0328 Low Dose Group | AZD0328 Optimal Dose Group | AZD0328 High Dose Group | Placebo
Number analyzed (Participants) | 23 | 32 | 13 | 19
units on a scale | 0.234 (0.122) [lower limit 0.122] | 0.240 (0.072) [lower limit 0.072] | 0.194 (0.216) [lower limit 0.216] | 0.266 (0.099) [lower limit 0.099]

2. Secondary Outcome: CogState Groton Maze Learning Task (GMLT) Standardized Change Score at Day 14
Description: GMLT score is defined as the -log10 transform of the sum of the number of errors made during GMLT trials. Mean GMLT score was calculated as the average of the 2 hour, 5 hour, and 8 hour scores. The GMLT standardized change score was calculated as the change from baseline in the mean GMLT score divided by the within subject standard deviation. Scale range from negative infinity (worst value) to positive infinity (best value).
Time Frame: Baseline and Day 14
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZD0328 Low Dose Group | AZD0328 Optimal Dose Group | AZD0328 High Dose Group | Placebo
Number analyzed (Participants) | 23 | 32 | 13 | 19
units on a scale | 0.313 (0.163) [lower limit 0.163] | 0.360 (0.104) [lower limit 0.104] | 0.281 (0.249) [lower limit 0.249] | 0.235 (0.124) [lower limit 0.124]

3. Secondary Outcome: CogState One Card Learning Task (OCLT) Standardized Change Score at Day 14
Description: OCLT score is defined as the arcsine transform of the proportion of correct responses during OCLT trials. Mean OCLT score was calculated as the average of the 2 hour, 5 hour, and 8 hour scores. The OCLT standardized change score was calculated as the change from baseline in the mean OCLT score divided by the within-subject standard deviation. Scale range from negative infinity (worst value) to positive infinity (best value).
Time Frame: Baseline and Day 14
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZD0328 Low Dose Group | AZD0328 Optimal Dose Group | AZD0328 High Dose Group | Placebo
Number analyzed (Participants) | 23 | 33 | 13 | 19
units on a scale | 0.150 (0.126) [lower limit 0.126] | 0.102 (0.100) [lower limit 0.100] | 0.094 (0.232) [lower limit 0.232] | 0.316 (0.152) [lower limit 0.152]

4. Secondary Outcome: CogState Detection Task (DT) Standardized Change Score at Day 14
Description: DT score is defined as -1 times the mean of log10 transformed reaction times for all correct responses. Mean DT score was calculated as the average of the 2 hour, 5 hour, and 8 hour scores. The DT standardized change score will be calculated as the change from baseline in the mean DT score divided by the within-subject standard deviation. Score range from negative infinity (worst value) to positive infinity (best value).
Time Frame: Baseline and Day 14
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZD0328 Low Dose Group | AZD0328 Optimal Dose Group | AZD0328 High Dose Group | Placebo
Number analyzed (Participants) | 23 | 33 | 13 | 19
units on a scale | 0.116 (0.116) [lower limit 0.116] | -0.014 (0.115) [lower limit 0.115] | -0.095 (0.158) [lower limit 0.158] | 0.098 (0.095) [lower limit 0.095]

5. Secondary Outcome: CogState Identification Task (IT) Standardized Change Score at Day 14
Description: IT score defined as 1 times the mean of log10 transformed reaction times for all correct responses. Mean IT score calculated as the average of the 2 hour, 5 hour, and 8 hour scores. The IT standardized change score will be calculated as the change from baseline in the mean IT score divided by the within-subject standard dev. Least square means were derived using a mixed effects repeated measures model with protocol scheduled assessment day, treatment group, baseline score, and assessment day-by-treatment interaction as fixed factors, center as a random factor, and baseline score as a covariate
Time Frame: Baseline and Day 14
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | AZD0328 Low Dose Group | AZD0328 Optimal Dose Group | AZD0328 High Dose Group | Placebo
Number analyzed (Participants) | 23 | 33 | 13 | 19
unit on a scale | -0.145 (0.177) [lower limit 0.177] | -0.049 (0.121) [lower limit 0.121] | -0.173 (0.136) [lower limit 0.136] | -0.103 (0.132) [lower limit 0.132]

6. Secondary Outcome: CogState Groton Maze Recall Task (GMRT) Standardized Change Score at Day 14
Description: GMRT score defined as the -log10 transform of the sum of the number of errors made during GMRT trials. Mean GMRT score calculated as the average of the 2 hour, 5 hour, and 8 hour scores. The GMRT standardized change score was calculated as change from baseline in mean GMRT score divided by the within subject standard deviation. Least square means were derived using a mixed effects repeated measures model with protocol scheduled assessment day, treatment group, baseline score, assessment day-by-treatment interaction as fixed factors, center as random factor, and baseline score as a covariate
Time Frame: Baseline and Day 14
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | AZD0328 Low Dose Group | AZD0328 Optimal Dose Group | AZD0328 High Dose Group | Placebo
Number analyzed (Participants) | 23 | 33 | 13 | 19
unit on a scale | 0.213 (0.139) [lower limit 0.139] | 0.406 (0.112) [lower limit 0.112] | 0.467 (0.263) [lower limit 0.263] | 0.409 (0.183) [lower limit 0.183]

ADVERSE EVENTS:
Arm/Group | AZD0328 Low Dose Group | AZD0328 Optimal Dose Group | AZD0328 High Dose Group | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/37 | 0/18 | 1/22
Other Adverse Events (participants affected / at risk) | 17/23 | 22/37 | 11/18 | 11/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0328 Low Dose Group (N=23) | AZD0328 Optimal Dose Group (N=37) | AZD0328 High Dose Group (N=18) | Placebo (N=22)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0328 Low Dose Group (N=23) | AZD0328 Optimal Dose Group (N=37) | AZD0328 High Dose Group (N=18) | Placebo (N=22)
DYSPEPSIA (Gastrointestinal disorders) | 9 | 10 | 5 | 4
HEADACHE (Nervous system disorders) | 6 | 4 | 6 | 4
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 2 | 4 | 0
CONSTIPATION (Gastrointestinal disorders) | 3 | 3 | 0 | 1
INSOMNIA (Psychiatric disorders) | 0 | 3 | 2 | 0
LETHARGY (Nervous system disorders) | 0 | 4 | 1 | 0
SEDATION (Nervous system disorders) | 1 | 2 | 2 | 1
ANXIETY (Psychiatric disorders) | 0 | 2 | 2 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 3 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication or presentation of results until the earlier of the publication of the first multi-center publication and the second anniversary of the completion of the multi-center study at all sites. Sponsor must receive a copy of proposed manuscript for review and comment at least 60 days prior to its submission for publication or presentation.